CLINICAL TRIAL: NCT00530309
Title: Clinical Assessment of GSK716155 for Type 2 Diabetes Mellitus -A Phase I/II Study to Investigate the Safety, Pharmacokinetics and Pharmacodynamics of GSK716155 in Japanese Subjects With Type 2 Diabetes Mellitus
Brief Title: Clinical Assessment of GSK716155 for Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: GLP107865
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GLP-1; type 2 diabeted mellitus; safety; GSK716155; GLP-1 receptor agonist; tolerability; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving GSK716155 + placebo (Experimental): Eligible subjects will receive GSK716155 with doses of 15 milligrams once a week, 30 milligrams once a week, 50 milligrams biweekly or 100 milligrams once every four weeks. Subjects will also receive placebo.
  Interventions: Drug: GSK716155 for injection; Drug: Placebo

INTERVENTIONS:
Drug: GSK716155 for injection — GSK716155 will be available with doses of 15 milligrams once a week, 30 milligrams once a week, 50 milligrams biweekly or 100 milligrams once every four weeks.
Drug: Placebo — Subjects will also receive placebo.

SUMMARY:
A Phase I/II study to investigate the safety, pharmacokinetics and pharmacodynamics of GSK716155 in Japanese subjects with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus diagnosed at least 3 months with FPG level <=240mg/dL and HbA1c between 6.5% and 10% inclusive.
* Must be diet controlled - OR - taking a single oral antidiabetic agent (other than thiazolidinediones) and willing to withdraw from this treatment from 2 weeks prior to the study.
* Must have a BMI:<=35kg/m2, 20 to 70 years of age inclusive.
* Woman must be of non-childbearing potential.

Exclusion criteria:

* Positive test result for either syphilis, HBs antigen, HCV antibody, HIV antigen/antibody, or HTLV-1 antibody.
* Clinically significant hepatic enzyme elevation.
* History of metabolic disease other than T2DM.
* Previous use of insulin as a treatment for diabetes within 3 months.
* History of severe gastrointestinal disease.
* Clinically significant cardiovascular disease.
* Significant renal disease as defined by screening lab test.
* History of drug (including albumin or albumin containing agents) allergy.
* History of alcohol or drug abuse.
* Donation of blood in excess of 400mL within previous 4 months.
* Previously received any GLP-1 mimetic or any other albumin-containing products.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2008-04-17 (Actual); Study Completion 2008-04-17 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations and PD parameters over time and at the end of study | Up to Week 9

SECONDARY OUTCOMES:
Other metabolic parameters at the end of study | Up to Week 9

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Seino Y, Nakajima H, Miyahara H, Kurita T, Bush MA, Yang F, Stewart MW. Safety, tolerability, pharmacokinetics and pharmacodynamics of albiglutide, a long-acting GLP-1-receptor agonist, in Japanese subjects with type 2 diabetes mellitus. Curr Med Res Opin. 2009 Dec;25(12):3049-57. doi: 10.1185/03007990903372999. PMID 19863477
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Results for study GLP107865 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/GLP107865?search=study&study_ids=GLP107865#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: GLP107865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: GLP107865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: GLP107865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: GLP107865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: GLP107865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: GLP107865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: GLP107865 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register